CLINICAL TRIAL: NCT01402154
Title: The Pre-treatment Detection of Circulating, Functional, Prostate Cells Among Adenocarcinoma Patients: an Evaluation of the EPISPOT Technique
Brief Title: EPISPOT Detection of Circulating Prostate Cells Among Adenocarcinoma Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOI/2010/SD-01; 2011-A00328-33 (Other: RCB number)
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Adenocarcinoma of the Prostate
MeSH Terms: interventions — Functional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Following the completion of the biological analyses required for this study, leftover tubes may be placed in the Nîmes University Hospital biological collection for future ancillary studies, if patients are agreed with this. The samples concerned include EDTA and CellSave tubes for each patient.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All study patients: All patients included according to stated inclusion and exclusion criteria.
  Interventions: Biological: EPISPOT detection of the number of circulating cells; Biological: CellSearch detection of the number of circulating, functional, prostate cells

INTERVENTIONS:
Biological: EPISPOT detection of the number of circulating cells — EPISPOT detection of the number of circulating, functional, prostate cells per unit blood
Biological: CellSearch detection of the number of circulating, functional, prostate cells — CellSearch detection of the number of circulating, functional, prostate cells per unit blood

SUMMARY:
The primary objective of this study is to evaluate the predictive value (in terms of remission) of a new technique for detecting circulating, functional, prostate cells among patients with localized adenocarcinoma of the prostate, and prior to any treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Histologically proven presence of prostate adenocarcinoma
* Localized disease on digital rectal examination
* Cancer without extensions
* Acceptance of a curative treatment by the patient

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is taking a hormone-modifying treatment
* Patient taking adrogenic supplements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically proven, localized, adenocarcinoma of the prostate who accept a curative treatment.
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2012-01-03 (Actual); Primary Completion 2014-12-08 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The difference between AUCs for the EPISPOT and Cellsearch Techniques | 1 day
  The difference between the AUCs (area under the curve) for the EPISPOT and Cellsearch techniques for detecting functional, circulating prostate cells

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Droupy, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (5):
- France (5):
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard
  - Clinique Beau Soleil, Montpellier
  - CHU de Montpellier - Hôpital Lapeyronie - Plateforme LCCRH, Montpellier
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier
  - Centre Regional de Lutte Contre le Cancer - Val d'Aurelle - Paul Lamarque, Montpellier